CLINICAL TRIAL: NCT02733315
Title: Long-term Effectiveness of the Diabetes Conversation Map Program: A Pre-post Education Intervention Study Among Diabetic Patients in Taiwan
Brief Title: Effectiveness of the Diabetes Conversation Map Program Among Diabetic Patients in Taiwan
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dalin Tzu Chi General Hospital (Other)
Responsible Party: Principal Investigator, Tzung-Yi Tsai, Assistant Researcher, Dalin Tzu Chi General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: DTCRD103-I-04
Record Dates: First submitted 2016-04-01; First posted 2016-04-11 (Estimated); Last update posted 2016-04-12 (Estimated); Status verified 2016-04

CONDITIONS: Diabetes
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- DCMP (Experimental)
  Interventions: Behavioral: Diabetes Conversation Map Program

INTERVENTIONS:
Behavioral: Diabetes Conversation Map Program — The experiment group received seven DCMP-based group education sessions for seven consecutive weeks in addition to routine health education at a private room in the outpatient unit. One registered nurse who received DCMP facilitator training, from the Taiwanese Association of Diabetic Educators, served as the class facilitator. DCMP sessions were conducted using seven colored "maps" covering different topics, including "walk with diabetes," "what is diabetes?", "a healthy diet and exercise," "walk with insulin," "diabetes complications and related risk factors," "foot care for diabetes patients," and "a type 1 diabetes patient in the home." Each map, a laminated 3-by-5-foot table-top visual with colorful drawings as metaphors of situations familiar to DM patients, was placed on a table with participants gathered around it. This procedure served to create mutual imagery to be shared with participants.

SUMMARY:
The Diabetes Conversation Map Program (DCMP) is a novel, group-based, interactive diabetes management education program that has been shown to help patients adapt to their disease. So the investigators aimed to examine the long-term effectiveness of the DCMP among diabetes patients in Taiwan.

DETAILED DESCRIPTION:
Study design and participants

A quasi-experimental pre-posttest control group design, with purposive sampling, was used to recruit participants from the Endocrinology department of a hospital in southern Taiwan from January to May of 2014. The inclusion criteria were (i) being at least 20 years old at the time of recruitment (ii) having no cognitive impairment and severe complications, (iii) being able to express opinions in either Mandarin or Taiwanese, and (iv) having a diagnosis of diabetes. To ensure participants' anonymity, all questionnaires were marked with an encryption code to facilitate data analysis, but with no personal identifiers.

Sample size calculation

Sample size calculation for this analysis of repeated measures to detect an effect size of 0.2 at 80% power and a 0.05 significance level indicated that a sample size of 68 patients is needed (according to G- POWER 3.1 analytical software, Franz Faul, Universitat Kiel, Germany). A sample of at least 89 participants for both groups combined was required on the basis of these parameters, allowing for a 30% attrition rate.

Intervention

Because continued participation was essential for this study, the participants were divided into the experiment or control group in accordance with the personal willingness. The control group received routine health education lasting for about 30 minutes per medical visit, which consisted of consultation about disease symptoms, related treatments, and self-care skills. They would receive health education instruction leaflets for reference purposes if necessary.

The experiment group received seven Diabetes Conversation Map Program (DCMP) -based group education sessions (10-12 participants, 1.5 hours each) for seven consecutive weeks in addition to routine health education at a private room in the outpatient unit. One registered nurse who received DCMP facilitator training, from the Taiwanese Association of Diabetic Educators, served as the class facilitator. DCMP sessions were conducted using seven colored "maps" covering different topics, including "walk with diabetes," "what is diabetes?", "a healthy diet and exercise," "walk with insulin," "diabetes complications and related risk factors," "foot care for diabetes patients," and "a type 1 diabetes patient in the home." Each map, a laminated 3-by-5-foot table-top visual with colorful drawings as metaphors of situations familiar to DM patients, was placed on a table with participants gathered around it. This procedure served to create mutual imagery to be shared with participants. In addition to using these colored maps, the facilitator further offered participants self-designed conversation cards and asked them to share individual glycemic control experiences based on the questions shown on the cards.

Outcome measures

The primary outcomes comprised the weekly self-monitoring of blood glucose (SMBG) times and some biochemical parameters containing BMI, HbA1c and fasting plasma glucose (FPG). In addition, the depressive symptoms as well as the level of diabetes health literacy were also measured, which were determined by the Taiwanese Depression Questionnaire (TDQ) and a self-administered questionnaire regarding diabetes health literacy.

The TDQ was developed according to the criteria specified by the Diagnostic and Statistical Manual of Mental Disorders (Third Edition) and consists of 18 self-reported items. Its total score ranged from 0 to 54, with higher scores indicating more severe depressive symptoms.

On the other hand, as to the diabetes health literacy, it was measured by a self-developed questionnaire. This scale contained 20 items and was scored using a 5-point Likert scale, with higher total scores indicating more positive diabetic health literacy.

Covariates Additional items addressing demographic and disease characteristics were developed based on clinical experience and literature review, and were collected at study entry via patient interviews and medical records. Demographic data included sex, age, marital status, education level, religion, household status, monthly income, and certain lifestyle factors, such as smoking, exercise habits, and presence of sleep disturbances. Smoking status was recorded as "non-smoker" or "current or ex-smoker." Those who exercised regularly (i.e., weekly) were classified as having "exercise habits." Sleep disturbances were defined as waking up at night more than twice without external factors during the week before the interview. Disease characteristics included the presence of chronic disease (i.e., stroke, hypertension, heart disease, renal disease, or cancer), medication regimen, and duration of diabetes.

Data collection procedure

The study protocol was approved by the Ethics Committee of Dalin Tzuchi Hospital (No. B10002009) prior to the recruitment of participants. Researchers explained the purpose of study and its procedure to all participants. Signed informed consent was obtained after they understood and agreed to participate in this study. Thereafter, investigators applied an observer-blind approach for data collection. A trained interviewer, who was not familiar with the participants, was assigned to collect the participants' information on demographic and disease characteristics. All data were obtained at three time points: before DCMP (T0), three days after DCMP (T1), and three months after DCMP (T2). To reduce the dropout rate, researchers asked participants to return the hospital for the completion of assessments via phone reminders. However, participants were still given the option to withdraw from the study at any time without any penalty.

Statistical analysis

Descriptive and inferential statistical analyses were conducted in accordance with the study aims and the nature of the variables. Descriptive parameters, including mean, standard deviation (SD), and percentage, were used to describe the distributions of demographic and disease data. Differences between the two groups were compared initially using t-test and χ2 test as appropriate. For inferential analysis, investigators used generalized estimating equation (GEE) procedure with identity link function with normal distribution to assess the long-term effects of DCMP, while taking into account within-subject correlations between measurements over time and the influence of potential confounding covariates. All analyses were conducted using SAS statistical software, Version 9.3. A p value of < .05 was considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* being at least 20 years old at the time of recruitment,
* having no cognitive impairment and severe complications,
* being able to express opinions in either Mandarin or Taiwanese, and
* having a diagnosis of DM.

Exclusion Criteria:

* being unwillingness to participant this work
* Attending the similar health education program in the past

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 95 (Actual)
Dates: Start 2014-01; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Weekly self-monitoring of blood glucose times as determined by medical chart review | Up to nine months

SECONDARY OUTCOMES:
Body mass index as determined by medical chart review | Up to nine months
The depressive symptoms level as measured by Taiwanese Depression Questionnaire | Up to nine months
Level of DM health literacy as measured by the self-developed questionnaire | Up to nine months
HbA1c as determined by medical chart review | Up to nine months
fasting plasma glucose as determined by medical chart review | Up to nine months

IPD SHARING:
Plan to Share IPD: Undecided